CLINICAL TRIAL: NCT05559073
Title: Outcomes of Early Referral to Radiofrequency Ablation in Symptomatic Atrial Fibrillation
Brief Title: Outcomes of Early Referral to Radiofrequency Ablation in Symptomatic Atrial Fibrillation Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Abdelrady Abdelsalam Farghaly, Assistant lecturer of cardiovascular medicine, Assiut University
Other Study IDs: Early Referral to AF Ablation
Record Dates: First submitted 2022-09-24; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation; Radiofrequency Ablation
Keywords: Early referral, catheter ablation, atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early referral to ablation within one year after first documented AF diagnosis
  Interventions: Procedure: Radiofrequency ablation
- Delayed referral to ablation after one year after first documented AF diagnosis
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — pulmonary vein isolation using radiofrequency ablation.

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia among adults with increasing risk of stroke, heart failure and mortality.

The EAST-AFNET 4 trial showed that rhythm control treatment (Antiarrhythmic drugs AAD or catheter ablation) was associated with a lower risk of adverse cardiovascular outcomes than usual care among patients who had recently (within one year) been diagnosed with atrial fibrillation.

In phase II/III GLORIA AF registry, Early AF ablation within 3 months from initial diagnosis in a contemporary cohort of patients who were predominantly treated with non-vitamin K antagonist oral anticoagulants was associated with a survival advantage compared to medical therapy alone.

Moreover, early AF ablation appeared to provide the greatest benefit compared to other treatments.

The ATTEST trial was a multicenter, randomized, prospective study in patients with paroxysmal atrial fibrillation (AF) designed to assess whether radiofrequency (RF) ablation is more effective in delaying the progression to persistent AF than AADs.

Patients >_65 years were significantly more likely to progress to persistent AF/AT than patients were <65 years, suggesting that early RF ablation may be an effective treatment strategy for delaying AF progression.

So, we hypothesize that early AF ablation within one year after first AF diagnosis may associate with improved procedures outcomes in symptomatic AF patients.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal and persistent atrial fibrillation (AF) documented on a 12 lead ECG, trans-telephonic monitoring (TTM) or Holter monitor (episodes of AF must be >30 seconds in duration to qualify as an inclusion criterion)
* Age of 18 years or older on the date of consent.
* Candidate for ablation based on AF that is symptomatic
* Informed Consent

Exclusion Criteria:

Permenant AF

* Previous left atrial (LA) ablation or LA surgery
* AF due to reversible cause (e.g. hyperthyroidism, cardiothoracic surgery)
* Active intracardiac thrombus
* Pre-existing pulmonary vein stenosis or pulmonary vein stent
* Contraindication to anticoagulation or radiocontrast materials
* Left atrial anteroposterior diameter greater than 5.5 cm by transthoracic echocardiography
* Cardiac valve prosthesis
* Severe mitral valve regurgitation or stenosis
* Myocardial infarction, percutaneous intervention, or coronary artery stenting during the 3-month period preceding the consent date
* Cardiac surgery during the three-month interval preceding the consent date
* Significant unrepaird congenital heart defect (including patent foramen ovale)
* NYHA class IV congestive heart failure
* Significant chronic kidney disease (eGFR <30 mL/min/1.73m2)
* Cerebral ischemic event (stroke or transient ischemic attack) during the six-month interval preceding the consent date
* Pregnancy and Life expectancy less than one year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We enroll all symptomatic AF patients who referred to first (de- novo) RF ablation within (early) vs. after (late) one year from the first AF diagnosis.
Sampling Method: Probability Sample
Enrollment: 127 (Estimated)
Dates: Start 2022-10-06 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from any atrial arrhythmia after single ablation procedure. | 12 months
  freedom from any documented atrial arrhythmia lasted for more than 30 seconds.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kuck KH, Lebedev DS, Mikhaylov EN, Romanov A, Geller L, Kalejs O, Neumann T, Davtyan K, On YK, Popov S, Bongiorni MG, Schluter M, Willems S, Ouyang F. Catheter ablation or medical therapy to delay progression of atrial fibrillation: the randomized controlled atrial fibrillation progression trial (ATTEST). Europace. 2021 Mar 8;23(3):362-369. doi: 10.1093/europace/euaa298. PMID 33330909